CLINICAL TRIAL: NCT04589988
Title: Building Capacity to Improve Community Participation for People Aging With Long-Term Disability Through Evidence-Based Strategies
Brief Title: Aging With Long Term Physical Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201710186
Record Dates: First submitted 2020-09-08; First posted 2020-10-19 (Actual); Results first posted 2024-11-18 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Physical Disability
Keywords: community participation; environmental modifications; home modifications; fall prevention

STUDY DESIGN:
Intervention Model Description: Parallel-group, randomized control, participants in the waitlist control group will receive the intervention after 6-month follow up is completed
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REBIL- Intervention arm (Experimental): Participants in this arm will receive the Removing Environmental Barriers to Independent Living (REBIL) intervention.
  Interventions: Behavioral: Removing Environmental Barriers to Independent Living (REBIL)
- Waitlist Attentional control (Other): Participants in this arm will receive life interview visits provided by a trained occupational therapist (OT) or OT student remotely for an equivalent amount of time to the treatment group. The waitlist control group will be offered the REBIL intervention after the 6-month follow-up is completed.
  Interventions: Behavioral: Waitlist Attentional Control

INTERVENTIONS:
Behavioral: Removing Environmental Barriers to Independent Living (REBIL) — REBIL is a complex intervention with two essential components: (1) removing environmental barriers and home hazards in the home tailored to the participant's unique abilities and limitations and (2) strategy training with the participant to help participant to be able to identify barriers in the home and community and identify potential resources and strategies to remove the barriers. Treatment includes one assessment session and four 75-minute visits in the home with an occupational therapist over 8 weeks, followed by a 6 -month assessment session by a blinded rater.
  Arms: REBIL- Intervention arm
Behavioral: Waitlist Attentional Control — The waitlist attentional control group will receive an initial assessment session then four 75 minute interview visits from an occupational therapy graduate assistant, followed by a 6-month assessment session by a blinded rater. After the 6-month follow-up is completed this group will receive the REBIL intervention.
  Arms: Waitlist Attentional control

SUMMARY:
The purpose of this study is to determine the feasibility and efficacy of an adapted evidence-based program (REBIL) to reduce barriers to community participation and remove fall hazards at home for adults aging with physical disabilities.

DETAILED DESCRIPTION:
Investigators will test the working hypothesis that the adapted program, focused on resolving environmental barriers, removing fall hazards, and building self-management skills in the home and community, will be feasible and superior to usual care for daily activity performance and participation outcomes in adults aging with physical disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-65 years
* Self-report of difficulty with at least 2 daily activities using the Older Adult Retirement Survey Activities of Daily Living (OARS ADL) scale
* onset of a physical disability 5 years prior to participation (e.g., spinal cord injury (SCI), cerebral palsy, post-polio syndrome, stroke, amputation).
* live within 60 miles of the research lab

Exclusion Criteria:

* Currently institutionalized.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Stark, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
The data (feasibility, primary and secondary outcomes) will be shared via a data repository.

REFERENCES:
- [Background] Chen SW, Somerville E, Devine M, Stark S. A protocol for Removing Environmental Barriers to Independent Living (REBIL): An adapted evidence-based occupational therapy intervention to increase community participation for individuals aging with long-term physical disabilities. Br J Occup Ther. 2022;86(5):349-58. doi: 10.1177/03080226221126901. PMID 38529197

RESULTS

PARTICIPANT FLOW:
Groups:
- REBIL- Intervention Arm: Participants in this arm received the Removing Environmental Barriers to Independent Living (REBIL) intervention.
  Removing Environmental Barriers to Independent Living (REBIL): REBIL is a complex intervention with two essential components: (1) removing environmental barriers and home hazards in the home tailored to the participant's unique abilities and limitations and (2) strategy training with the participant to help participant to be able to identify barriers in the home and community and identify potential resources and strategies to remove the barriers. Treatment includes one assessment session and four 75-minute visits in the home with an occupational therapist over 8 weeks, followed by a 6 -month assessment session by a blinded rater.
- Waitlist Attentional Control: Participants in this arm were received life interview visits provided by a trained occupational therapist (OT) or OT student remotely for an equivalent amount of time to the treatment group. The waitlist control group will be offered the REBIL intervention after the 6-month follow-up is completed.
  Waitlist Attentional Control: The waitlist attentional control group will receive an initial assessment session then four 75 minute interview visits from an occupational therapy graduate assistant, followed by a 6-month assessment session by a blinded rater. After the 6-month follow-up is completed this group will receive the REBIL intervention.
Period: Overall Study
Arm/Group | REBIL- Intervention Arm | Waitlist Attentional Control
Started | 24 | 26
Completed | 23 | 24
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | REBIL- Intervention Arm | Waitlist Attentional Control | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (4.4) | 58.4 (5.3) | 57.8 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 8 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and ethnicity: Black/African American | 9 | 8 | 17
  Race and ethnicity: Hispanic or Latino | 1 | 0 | 1
  Race and ethnicity: White | 13 | 16 | 29
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47
Living situation [Count of Participants; unit: Participants]
  Lives with someone | 13 | 14 | 27
  Lives alone | 10 | 10 | 20
Receives assistance with daily activities [Count of Participants; unit: Participants]
  Yes | 14 | 14 | 28
  No | 9 | 10 | 19
Work status [Count of Participants; unit: Participants]
  Working full-time/part-time | 6 | 7 | 13
  Disability leave | 12 | 15 | 27
  Retired/other | 5 | 2 | 7
Use of mobility device [Count of Participants; unit: Participants]
  None | 3 | 2 | 5
  Wheelchair | 6 | 9 | 15
  Other device (e.g., cane, walker) | 14 | 13 | 27
PROMIS Depression [Mean (Standard Deviation); unit: T-score] — Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Scale-Short Form 8-item. Uncorrected t-scores were calculated by the PROMIS scoring system, with higher scores indicating higher level of depressive symptoms. A score of 50 is the average of the US general population, with a standard deviation of 10.
  T-score | 53.5 (9.6) | 54.6 (9.0) | 54.1 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: In-Home Occupational Performance Evaluation (I-HOPE) Activity Score
Description: The In-Home Occupational Performance Evaluation (I-HOPE) activity score measures current activity patterns of participants across 44 activities. The score ranges from 0 to 1.0, with a higher score indicating fewer problematic activities for the participant.
Time Frame: Baseline and 6-month follow up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REBIL- Intervention Arm | Waitlist Attentional Control
Number analyzed (Participants) | 23 | 24
score on a scale
  Baseline | 0.73 (0.03) | 0.72 (0.03)
  6-month follow up | 0.76 (0.03) | 0.69 (0.03)
Statistical Analysis 1: Comparison: REBIL- Intervention Arm vs Waitlist Attentional Control; A linear mixed effects model was used to assess the effects of time (6-month follow-up versus baseline), group (REBIL versus control) and the interaction of group and time on the outcome. A significant interaction of group and time would indicate that the two groups had significantly different changes in the outcome over time. The model adjusted for age, sex, race, and depression score at baseline; Test type: Superiority; p = 0.068, Mixed Models Analysis — P value shown is for group by time interaction

2. Primary Outcome: In-Home Occupational Performance Evaluation (I-HOPE) Performance Score
Description: The In-Home Occupational Performance Evaluation (I-HOPE) performance score is a mean rating across up to 10 participant-prioritized activities on a scale of 1 (unable to perform the activity at all) to 5 (able to perform the activity without difficulty).
Time Frame: Baseline and 6-month follow up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REBIL- Intervention Arm | Waitlist Attentional Control
Number analyzed (Participants) | 23 | 24
score on a scale
  Baseline | 2.49 (0.15) | 2.52 (0.15)
  6-month follow up | 3.23 (0.15) | 2.87 (0.15)
Statistical Analysis 1: Comparison: REBIL- Intervention Arm vs Waitlist Attentional Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.063, Mixed Models Analysis — P value shown is for group by time interaction

3. Primary Outcome: In-Home Occupational Performance Evaluation (I-HOPE) Satisfaction Score
Description: The In-Home Occupational Performance Evaluation (I-HOPE) satisfaction score is a mean rating across up to 10 participant-prioritized activities on a scale of 1 (not satisfied at all with the performance of the activity) to 5 (very satisfied with their performance of the activity).
Time Frame: Baseline and 6-month follow up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REBIL- Intervention Arm | Waitlist Attentional Control
Number analyzed (Participants) | 23 | 24
score on a scale
  Baseline | 2.12 (0.17) | 2.09 (0.18)
  6-month follow-up | 2.86 (0.17) | 2.74 (0.18)
Statistical Analysis 1: Comparison: REBIL- Intervention Arm vs Waitlist Attentional Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.724, Mixed Models Analysis — P value shown is for group by time interaction

4. Primary Outcome: In-Home Occupational Performance Evaluation (I-HOPE) Barrier Severity Score
Description: The In-Home Occupational Performance Evaluation (I-HOPE) barrier severity score is a total sum of barrier ratings (0=independent with/without a device, 1=stand-by assistance needed, 2=minimum assistance needed, 3=moderate assistance needed, 4=maximum assistance needed, 5=no activity) for all identified barriers across up to 10 prioritized activities. Multiple barriers could be identified for each prioritized activity. Higher scores indicate greater barrier severity. There is no maximum score.
Time Frame: Baseline and 6-month follow up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REBIL- Intervention Arm | Waitlist Attentional Control
Number analyzed (Participants) | 23 | 24
score on a scale
  Baseline | 50.28 (4.78) | 51.83 (4.82)
  6-month follow up27.79 | 21.93 (4.78) | 27.79 (4.82)
Statistical Analysis 1: Comparison: REBIL- Intervention Arm vs Waitlist Attentional Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.447, Mixed Models Analysis — P value shown is for group by time interaction

5. Primary Outcome: Reintegration to Normal Living Index (RNLI)
Description: The Reintegration to Normal Living Index is a disability-related quality-of life-instrument that will be used to measure participants' satisfaction with their home and community participation and has been validated on a population of community-dwelling individuals with chronic conditions. It uses an 11-item, 10 point visual analog scale with higher scores indicating greater reintegration to normal living. The sum score is divided by 110 and then multiplied by 100 to obtain an adjusted score. Adjusted scores range from 0 to 100, with higher scores indicating greater reintegration to normal living.
Time Frame: Baseline and 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REBIL- Intervention Arm | Waitlist Attentional Control
Number analyzed (Participants) | 23 | 24
score on a scale
  Baseline | 65.59 (3.56) | 66.10 (3.72)
  6-month follow up | 70.08 (3.52) | 68.90 (3.72)
Statistical Analysis 1: Comparison: REBIL- Intervention Arm vs Waitlist Attentional Control; A linear mixed effects model was used to assess the effects of time (6-month follow-up versus baseline), group (REBIL versus control) and the interaction of group and time on the outcome. A significant interaction of group and time would indicate that the two groups had significantly different changes in the outcome over time. The model adjusted for age, sex, race, work status, and depression score at baseline; Test type: Superiority; p = 0.696, Mixed Models Analysis — P value shown is for group by time interaction

6. Primary Outcome: Westmead Home Safety Assessment (WeHSA) Short Form
Description: The Westmead Home Safety Assessment (WeHSA) short form is a performance-based assessment of fall hazards in different spaces of the home (e.g., kitchen, bathroom, hallway, bedroom etc.). WeSHA scores indicate the total number of environmental fall hazards in the home.
Time Frame: Baseline and 6-month follow up
Measure: Least Squares Mean (Standard Error); unit: number of fall hazards
Arm/Group | REBIL- Intervention Arm | Waitlist Attentional Control
Number analyzed (Participants) | 23 | 24
number of fall hazards
  Baseline | 10.52 (1.05) | 9.94 (1.05)
  6-month follow up | 7.04 (1.05) | 6.94 (1.05)
Statistical Analysis 1: Comparison: REBIL- Intervention Arm vs Waitlist Attentional Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.798, Mixed Models Analysis — P value shown is for group by time interaction

7. Secondary Outcome: Fall Prevention Strategy Survey (FPSS)
Description: The Fall Prevention Strategy Survey is a self-report instrument addressing protective behaviors related to fall risk among adults. It is an 11-item survey, scores range from 0 to 22 with higher scores indicating use of more fall prevention strategies.
Time Frame: Baseline and 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | REBIL- Intervention Arm | Waitlist Attentional Control
Number analyzed (Participants) | 23 | 24
score on a scale
  Baseline | 13.2 (0.9) | 13.9 (0.9)
  6-month follow up | 16.5 (0.9) | 15.2 (0.9)
Statistical Analysis 1: Comparison: REBIL- Intervention Arm vs Waitlist Attentional Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.135, Mixed Models Analysis — P value shown is for group by time interaction

8. Secondary Outcome: Participation Scale
Description: This scale comprises 25 diverse activities across four participation domains: routines, recreation, responsibilities, and relationships. Ratings were on a five-point Likert-type scale regarding the frequency of participation, the importance of the activity, and their self-efficacy in completing it. We calculated the ratio of number of important/very important activities they could perform very much/as much as they wanted (numerator) to the number of important/very important activities (denominator).
Time Frame: Baseline and 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | REBIL- Intervention Arm | Waitlist Attentional Control
Number analyzed (Participants) | 23 | 24
ratio
  Baseline | 0.54 (0.05) | 0.58 (0.05)
  6-month follow-up | 0.65 (0.05) | 0.63 (0.05)
Statistical Analysis 1: Comparison: REBIL- Intervention Arm vs Waitlist Attentional Control; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.291, Mixed Models Analysis — P value shown is for group by time interaction

9. Secondary Outcome: Fall Rate
Description: Participants reported monthly on the number of falls they experienced in the past month. A fall was defined as an unexpected event in which a person comes to rest on the ground, floor, or a lower level. Fall rates were calculated as the number of falls per 1000 observed participant days.
Time Frame: 6 months
Measure: Number; unit: Rate of falls per 1000 participant days
Arm/Group | REBIL- Intervention Arm | Waitlist Attentional Control
Number analyzed (Participants) | 23 | 24
Rate of falls per 1000 participant days | 15 | 17.6
Statistical Analysis 1: Comparison: REBIL- Intervention Arm vs Waitlist Attentional Control; Fall rates were compared between REBIL and control groups using negative binomial regression. The model adjusted for age, sex, ace, and depression score at baseline. The null hypothesis was that fall rates do not differ between groups; Test type: Superiority; p = 0.631, Negative binomial regression; Incidence rate ratio = 0.83, 95% CI 2-sided [0.40 to 1.76] — IRR reflects REBIL intervention group versus control group

ADVERSE EVENTS:
Time Frame: 6 months from baseline
Arm/Group | REBIL- Intervention Arm | Waitlist Attentional Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT04589988/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT04589988/ICF_001.pdf